CLINICAL TRIAL: NCT06281626
Title: Use of the Free Male Condom Scheme in Young Adults Aged 18 to 25
Acronym: Préservatif
Status: Completed | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2024_RIPH_01_Preservatif
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-02

CONDITIONS: Comdom
Keywords: Young adults; condom; free condom; use of condom
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults: people aged 18 to 25 years.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
For several years, the incidence of sexually transmitted infections (STIs) has been rising sharply, while that of HIV has stagnated. This is due to the decline in condom use since the late 1990s, despite the fact that condom are considered the only effective way to prevent STIs.

In France, 40% of STIs concern young people aged 15 to 25. The national public health strategy aims to stem the circulation of HIV and eliminate STIs as a major public health problem by 2030. To achieve this, several measures have been implemented: reimbursement of male condoms on prescription (2018), 100% free contraception and prevention in sexual health consultation (2021), and more recently, free, non-prescription access to male condoms in pharmacies (end 2022).

DETAILED DESCRIPTION:
The main objective is to describe the use of free male condoms by young adults aged 18 to 25.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 25 years
* Male or female
* Regardless of their sexual orientation
* Agreeing to participate in the study

Exclusion Criteria:

* Minors
* Refusing to participate in the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People aged 18 to 25 years.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
use of free male condoms | Day 0
  use of free male condoms recorded as yes or not

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided